CLINICAL TRIAL: NCT01024816
Title: Practicing Restorative Yoga or Stretching for the Metabolic Syndrome
Acronym: PRYSMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01AT004569-01A2 (NIH)
Record Dates: First submitted 2009-12-01; First posted 2009-12-03 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic Syndrome; Restorative Yoga; Stretching; Visceral adiposity; Randomized controlled trial
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Restorative yoga intervention (Experimental)
  Interventions: Behavioral: Restorative yoga
- Stretching group (Active Comparator)
  Interventions: Behavioral: Stretching

INTERVENTIONS:
Behavioral: Restorative yoga — Group yoga sessions: Participants will attend 90 minute yoga group classes for 48 weeks: twice a week for 6 weeks, then once weekly during weeks 7 to 12, then every other week for weeks 13 - 24, and once a month for 6 months. We plan a progressive series of classes, with a subset of poses for each class and then selecting individual poses to focus on in each class.
  Home yoga practice: Participants will be given a video disk (DVD) of the yoga postures at the start of the yoga intervention practice. We will also provide the yoga participants with a written manual with pictures and descriptions of each posture that they will be taught in the group sessions. The participants will be asked to practice the postures taught during their group sessions at home at least three times a week with the assistance of the DVD and manual. Each participant will be given a set of yoga props for their use at home. We will ask all participants to keep a log of their home practice sessions
  Arms: Restorative yoga intervention
Behavioral: Stretching — Group classes: Participants will attend 90 minute group stretching classes for 48 weeks: twice a week for 6 weeks, then once weekly during weeks 7 to 12, then every other week for weeks 13 - 24, and once a month for 6 months. The stretches will address all body parts, including cervical, upper extremity, thoracic, lumbar, pelvic, and lower extremity musculature.
  Home stretching practice: Each participant will receive a written manual with pictures and descriptions of each stretch that they will be learning in group sessions and a DVD with instruction on each of the stretches. The participants will be asked to practice the stretches taught during their group sessions at home at least three times a week with the assistance of the DVD and manual. Each participant will be given stretching supplies. We will ask all participants to keep a log of their home practice sessions.
  Arms: Stretching group

SUMMARY:
The purpose of this study is to determine whether Restorative yoga versus stretching exercises will reduce risk factors for metabolic syndrome in adults with metabolic syndrome.

DETAILED DESCRIPTION:
Metabolic abnormalities, including visceral adiposity, insulin resistance, hyperglycemia, hypertension and dyslipidemia, occur together and are associated with excessive caloric intake and inadequate physical activity. Persons with the metabolic syndrome are at high risk of developing type 2 diabetes and cardiovascular disease. Lifestyle and behavioral interventions reduce these risks, but many individuals with increased metabolic risk find it difficult to achieve and maintain weight loss and increased physical activity.

We are conducting a rigorous randomized controlled trial at two clinical sites to determine if Restorative yoga compared to stretching exercises improves the metabolic syndrome among overweight and underactive individuals who meet criteria for the metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Anyone between the ages of 21 and 65 who may meet the criteria for the metabolic syndrome can sign-up for the screening process. A more thorough screening process will be conducted to determine whether or not you are eligible to enroll in the study
* Underactive
* Overweight

Exclusion Criteria:

* Pregnancy or breast feeding
* Chronic illnesses: cancer, kidney disease, cirrhosis of the liver, rheumatologic diseases, or chronic infections
* Not ambulatory or neurological condition causing impaired mobility
* Weight over 400 pounds
* History of or plans for bariatric surgery
* Inability to speak and read English

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2009-12; Primary Completion 2012-07 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
visceral adiposity by abdominal CT scan | 6-months and 12-months

SECONDARY OUTCOMES:
systolic blood pressure, fasting triglycerides, and fasting insulin levels (co-primary outcomes); change in glucose tolerance, HbA1c levels, high density lipoprotein (HDL) cholesterol, and quality of life (secondary outcomes). | 6-months and 12-months

CONTACTS AND LOCATIONS:
Overall Officials: Alka Kanaya, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, San Diego, San Diego, California
  - Unversity of California, San Francisco, San Francisco, California

REFERENCES:
- [Derived] Flowers E, Allen IE, Kanaya AM, Aouizerat BE. Circulating MicroRNAs predict glycemic improvement and response to a behavioral intervention. Biomark Res. 2021 Aug 23;9(1):65. doi: 10.1186/s40364-021-00317-5. PMID 34425916
- [Derived] Corey SM, Epel E, Schembri M, Pawlowsky SB, Cole RJ, Araneta MR, Barrett-Connor E, Kanaya AM. Effect of restorative yoga vs. stretching on diurnal cortisol dynamics and psychosocial outcomes in individuals with the metabolic syndrome: the PRYSMS randomized controlled trial. Psychoneuroendocrinology. 2014 Nov;49:260-71. doi: 10.1016/j.psyneuen.2014.07.012. Epub 2014 Jul 21. PMID 25127084
- See also: Related Info — http://coe.ucsf.edu/scor/prysms/